CLINICAL TRIAL: NCT06146738
Title: The PALSUR-study: Palliative Care Versus Surgery in High-grade Glioma Patients (ENCRAM 2203)
Acronym: PALSUR
Status: Recruiting | Type: Observational
Sponsor: Jasper Gerritsen (Other)
Collaborators: Haaglanden Medical Centre (Other); Universitaire Ziekenhuizen KU Leuven (Other); University Hospital Heidelberg (Other); Technical University of Munich (Other); Insel Gruppe AG, University Hospital Bern (Other); Massachusetts General Hospital (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor-Investigator, Jasper Gerritsen, Jasper K.W. Gerritsen MD PhD, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: MEC-2020-0812-4
Record Dates: First submitted 2023-11-18; First posted 2023-11-27 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioblastoma, IDH-wildtype; Glioblastoma Multiforme, Adult
Keywords: Palliative care; Best supportive care; Biopsy; Resection; Quality of life; Survival; Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Palliative Care; Transurethral Resection of Bladder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Palliative Care: Best supportive care without surgical intervention
  Interventions: Behavioral: Palliative Care
- Tumor biopsy: Tumor biopsy
  Interventions: Procedure: Tumor biopsy
- Tumor resection: Maximal safe resection of the tumor
  Interventions: Procedure: Tumor resection

INTERVENTIONS:
Behavioral: Palliative Care — Best supportive care without surgical intervention
  Other Names: Best Supportive Care
  Groups: Palliative Care
Procedure: Tumor biopsy — Tumor biopsy
  Groups: Tumor biopsy
Procedure: Tumor resection — Maximal safe resection of the tumor
  Groups: Tumor resection

SUMMARY:
There is no consensus on the optimal treatment of patients with high-grade glioma, especially when patients have limited functioning performance at presentation (KPS ≤70). Therefore, there are varied practice patterns around pursuing biopsy, resection, or palliation (best supportive care). This study aims to characterize the impact of palliative care versus biopsy versus resection on survival and quality of life in these patients. Also, it will aim to determine if there is a subset of patients that benefit the most from resection or biopsy, for which outcome, and how they could be identified preoperatively.

This study is an international, multicenter, prospective, 3-arm cohort study of observational nature. Consecutive HGG patients will be treated with palliative care, biopsy, or resection at a 1:3:3 ratio. Primary endpoints are: 1) overall survival, and 2) quality of life at 6 weeks, 3 months and 6 months after initial presentation based on the EQ-5D, EORTC QLQ C30 and EORTC BN 20 questionnaires. Total duration of the study is 5 years. Patient inclusion is 4 years, follow-up is 1 year.

DETAILED DESCRIPTION:
Trial design This is an international, multicenter, prospective, observational, 3-arm cohort study (registration: clinicaltrials.gov ID number TBA). Eligible patients are treated with either palliative care, biopsy, or resection with a 1:3:3 ratio with a sequential computer-generated random number as subject ID.

Study objectives The primary study objective is to evaluate safety and efficacy of palliative care versus surgery in HGG patients as measured by overall survival (OS) and quality of life questionnaires (QLQ C30, EORTC QLQ BN20, EQ 5D).

The primary outcomes are 1) overall survival (OS) defined as time from diagnosis to death from any cause; 2) proportion of patients with health-related quality of life deterioration of 10 points or more in the EORTC QLQ C30 questionnaire or EORTC QLQ BN20 questionnaire at 3 months after outpatient clinic visit.

Study setting and participants Patients will be recruited from the neurosurgical or neurological outpatient clinic or through referral from general hospitals of the participating neurosurgical hospitals, located in Europe and the United States. The study is carried out by centers from the ENCRAM Consortium.

Study patients are allocated to either the supramaximal or maximum safe resection group and will undergo evaluation at presentation (baseline) and during the follow-up period at 6 weeks, 3 months, and 6 months. Patient functioning with be assessed with the Karnofsky Performance Scale (KPS) and the ASA (American Society of Anesthesiologists) physical status classification system. Health-related quality of life (HRQoL) will be assessed with the EORTC QLQ C30, EORTC QLQ BN20 and EQ 5D questionnaires. Overall survival will be assessed at 6 months postoperatively. We expect to complete patient inclusion in 4 years. The estimated duration of the study (including follow-up) will be 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤90 years
2. Tumor diagnosed as HGG (WHO grade III/IV) on MRI as assessed by the neurosurgeon
3. Written informed consent

Exclusion Criteria:

1. Tumors of the cerebellum, brainstem or midline
2. Inability to give written informed consent
3. Secondary high-grade glioma due to malignant transformation from low-grade glioma
4. Second primary malignancy within the past 5 years with the exception of adequately treated in situ carcinoma of any organ or basal cell carcinoma of the skin

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the neurosurgical or neurological outpatient clinic or through referral from general hospitals of the participating neurosurgical hospitals, located in Europe and the United States. The study is carried out by centers from the ENCRAM Consortium.
Sampling Method: Non-Probability Sample
Enrollment: 1015 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | Up to 5 years postoperatively
  Time from diagnosis to death from any cause
Quality of life at 3 months (EORTC QLQ C30) | 3 months postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 3 months (EORTC QLQ BN20) | 3 months postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 3 months (EQ-5D) | 3 months postoperatively
  Quality of life as assessed by the EQ-5D questionnaire

SECONDARY OUTCOMES:
Quality of life at 6 weeks (EORTC QLQ C30) | 6 weeks postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 6 weeks (EORTC QLQ BN20) | 6 weeks postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 6 weeks (EQ-5D) | 6 weeks postoperatively
  Quality of life as assessed by the EQ-5D questionnaire
Quality of life at 6 months (EORTC QLQ C30) | 6 months postoperatively
  Quality of life as assessed by the EORTC QLQ C30 questionnaire
Quality of life at 6 months (EORTC QLQ BN20) | 6 months postoperatively
  Quality of life as assessed by the EORTC QLQ BN20 questionnaire
Quality of life at 6 months (EQ-5D) | 6 months postoperatively
  Quality of life as assessed by the EQ-5D questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Jasper Gerritsen, MD PhD, Principal Investigator — Erasmus Medical Center
Locations (8):
- United States (2):
  - University of California, San Francisco, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
- University Hospital Leuven, Leuven, Belgium
- Germany (2):
  - Technical University Munich, Munich, Bavaria
  - University Hospital Heidelberg, Heidelberg
- Netherlands (2):
  - Erasmus Medical Center, Rotterdam, South Holland
  - Haaglanden Medical Centre, The Hague, South Holland
- Inselspital Universitätsspital Bern, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided